CLINICAL TRIAL: NCT07105839
Title: A Prospective, Randomized Controlled Trial Comparing Opioid-Free and Opioid-Based Anesthesia in Morbidly Obese Patients Undergoing Bariatric Surgery
Brief Title: Opioid-Free Versus Opioid-Based Anesthesia in Bariatric
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Siirt Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, ali kendal oğuz, Specialist Doctor In Anestesiology And Reanimation, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OBES-OFAN-2025-01
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Bariatric Surgery
Keywords: Opioid-Free Anesthesia; Pain Management; Multimodal Analgesia; Quality of Recovery (QoR-15); TAP Block
MeSH Terms: conditions — Obesity; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group O (Opioid Group) (Active Comparator): Induction with: 2 mg/kg IV propofol, 2 μg/kg fentanyl, 0.6 mg/kg rocuronium (ideal body weight)
  Maintenance:0.1-0.3 μg/kg/min IV remifentanil infusion and 1 MAC sevoflurane
  Bilateral TAP block: 40 mL of 0.25% bupivacaine under ultrasound guidance
  Interventions: Drug: Intraoperative rescue analgesia
- Group NO (Opioid-Free Group) (Active Comparator): Induction with: 2 mg/kg IV propofol, 0.5 mg/kg ketamine, 0.6 mg/kg rocuronium
  Maintenance: 0.2-1.4 μg/kg/h IV dexmedetomidine and 1 MAC sevoflurane
  Bilateral TAP block: 40 mL of 0.25% bupivacaine under ultrasound guidance
  Interventions: Drug: Intraoperative rescue analgesia:

INTERVENTIONS:
Drug: Intraoperative rescue analgesia — If signs of inadequate analgesia occur (e.g., >20% increase in heart rate or blood pressure), IV remifentanil infusion rate will be titrated upward within the safety margin.
  Arms: Group O (Opioid Group)
Drug: Intraoperative rescue analgesia: — If signs of inadequate analgesia occur (e.g., >20% increase in heart rate or blood pressure), IV dexmedetomidine infusion rate will be titrated upward (up to maximum safe dose).
  Arms: Group NO (Opioid-Free Group)

SUMMARY:
This study is designed as a prospective, randomized, controlled clinical trial. It will be conducted in the operating rooms of the University of Health Sciences, Diyarbakır Gazi Yaşargil Training and Research Hospital. Patients aged 18 to 65 years who are scheduled for elective bariatric surgery and meet the inclusion criteria (ASA physical status I-III) will be enrolled in the study.

Eligible patients will be informed both verbally and in writing during their preoperative anesthetic evaluation, and written informed consent will be obtained at least 24 hours prior to surgery.

Patients will be randomly assigned to one of two groups using computer-generated randomization:

Group O (Opioid group)

Group NO (Opioid-free group)

All patients will receive 40 mg IV pantoprazole and 4 mg IV ondansetron 30 minutes before surgery as preoperative medication. Standard ASA monitoring will be applied, and fasting guidelines will be followed. Depth of anesthesia will be monitored in all patients using BIS, and maintained within a target range of BIS 40-60 to ensure adequate depth with no response to surgical stimuli.

DETAILED DESCRIPTION:
This study is designed as a prospective, randomized, controlled clinical trial. It will be conducted in the operating rooms of the University of Health Sciences, Diyarbakır Gazi Yaşargil Training and Research Hospital. Patients aged 18 to 65 years who are scheduled for elective bariatric surgery and meet the inclusion criteria (ASA physical status I-III) will be enrolled in the study.

Eligible patients will be informed both verbally and in writing during their preoperative anesthetic evaluation, and written informed consent will be obtained at least 24 hours prior to surgery.

Patients will be randomly assigned to one of two groups using computer-generated randomization:

Group O (Opioid group)

Group NO (Opioid-free group)

All patients will receive 40 mg IV pantoprazole and 4 mg IV ondansetron 30 minutes before surgery as preoperative medication. Standard ASA monitoring will be applied, and fasting guidelines will be followed. Depth of anesthesia will be monitored in all patients using BIS, and maintained within a target range of BIS 40-60 to ensure adequate depth with no response to surgical stimuli.

Anesthesia Protocol:

Group O (Opioid Group):

General anesthesia will be induced with 2 mg/kg propofol, 2 µg/kg fentanyl, and 0.6 mg/kg rocuronium based on ideal body weight (IBW). Maintenance will be achieved using remifentanil (Ultiva®) infusion at 0.1-0.3 µg/kg/min and 1 MAC sevoflurane. Following induction, all patients will receive a bilateral transversus abdominis plane (TAP) block under ultrasound guidance using 40 mL of 0.25% bupivacaine.

Group NO (Opioid-Free Group):

General anesthesia will be induced with 2 mg/kg propofol, 0.5 mg/kg ketamine, and 0.6 mg/kg rocuronium (IBW). Anesthesia will be maintained with dexmedetomidine infusion at 0.2-1.4 µg/kg/h and 1 MAC sevoflurane. Following induction, a bilateral TAP block will also be performed using 40 mL of 0.25% bupivacaine under ultrasound guidance.

Postoperative Analgesia Protocol:

During skin closure, all patients will receive 1 g IV paracetamol and 50 mg IV ketoprofen. At the end of surgery, neuromuscular blockade will be reversed using sugammadex, and patients will be safely extubated.

In the postoperative period, patients will be followed in the surgical ward for 48 hours with a standardized analgesic protocol:

1 g IV paracetamol every 6 hours

4 mg IV ondansetron every 8 hours

50 mg IV ketoprofen every 12 hours

Pain will be assessed using the Visual Analog Scale (VAS). If VAS ≥ 4, 100 mg IV tramadol will be administered as rescue analgesia, and all interventions will be documented in the patient records.

ELIGIBILITY:
Inclusion Criteria:

Age 18-65 years

BMI >35

ASA class III-IV

Elective bariatric surgery (e.g., sleeve gastrectomy)

Written informed consent

Exclusion Criteria:

Refusal to participate

Severe cardiac/pulmonary/psychiatric illness

Allergy to study drugs

Conversion to emergency surgery

Withdrawal at any point by patient or investigator

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative VAS pain scores | post-op 1.hour (H), 2.H, 3.H, 6.H, 12.H, 18.H, 24.H, 36.H and 48.H
QoR-15 score (Quality of Recovery) | 24 Hours and 48 Hours

SECONDARY OUTCOMES:
Rescue analgesic requirement | Within 48 hours post-op
  IV tramadol
Postoperative nausea and vomiting (PONV) incidence questionnaire | 48 hours

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing is currently under consideration. A final decision will be made after study completion and ethical approval.